CLINICAL TRIAL: NCT01274988
Title: Deep Brain Stimulation of Nucleus Accumbens as a New Treatment to Prevent Relapse for Opiate Addicts
Brief Title: Deep Brain Stimulation of Nucleus Accumbens to Prevent Opiate Relapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Guodong Gao, Department of Neurosurgery, Tang-Du Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NACDBS
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Addiction
Keywords: Opiate dependence; Deep brain stimulation; Nucleus accumbens
MeSH Terms: conditions — Behavior, Addictive; Opioid-Related Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Experimental): Continuous deep brain stimulation of bilateral nucleus accumbens
  Interventions: Procedure: Deep brain stimulation
- Standard Control (Active Comparator): methadone maintenance treatment
  Interventions: Other: methadone maintenance treatment

INTERVENTIONS:
Procedure: Deep brain stimulation — Deep brain stimulation of bilateral nucleus accumbens
  Arms: Deep Brain Stimulation
Other: methadone maintenance treatment — methadone maintenance treatment
  Arms: Standard Control

SUMMARY:
Nucleus accumbens plays important roles in the process of opiate addiction and initial of relapse after detoxification, deep brain stimulation of nucleus accumbens will inhibit its activity and thus to effectively prevent the relapse of the opiate dependence.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Long lasting heroin addiction (fulfilled diagnostic-criteria according to ICD-10)
* At least three detoxication-treatments without a long-term period of abstinence has already taken place
* Long-term inpatient treatment to support abstinence have occurred
* completion of detoxification treatment preoperatively with no somatic symptoms of withdrawal
* negative morphine urinalysis and naloxone tests
* Free patient's decision/informed Consent (existing comprehensive ability in meaning, methodology and execution of the study and ability of acceptance)

Exclusion Criteria:

* Clinical relevant psychiatric comorbidity (schizophrenic psychoses, bipolar affective diseases, severe personality disorder)
* Contraindications of a MRI-examination, e.g. implanted cardiac pacemaker/heart defibrillator
* Current and in the last six months existent paranoid-hallucinated symptomatology
* Foreign aggressiveness in the last six months
* Stereotactic respectively neurosurgical intervention in the past
* Contraindications of a stereotactic operation, e.g. increased bleeding-disposition, cerebrovascular diseases (e.g. arteriovenous malfunction, aneurysms, systemic vascular diseases)
* Serious and instable organic diseases (e.g. instable coronal heart disease)
* tested positively for HIV
* pregnancy and/or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Treatment retention | 12 months
  Opiate abstinent time by self-reports and monthly urinalysis for the patients undergo the deep brain stimulation of nucleus accumbens,treatment retention time for the methadone maintenance treatment patients

SECONDARY OUTCOMES:
Change of participants' craving for opioid drugs | Baseline, 3 month, 6 month and 12month follow-up assessments
  The 10-point visual analog scale (VAS),will be utilized at each time point. A participants' diary will be utilized at each time point.
Change in Addiction Severity Index (ASI lite) composite scores | Baseline, 3 month, 6 month and 12month follow-up assessments
Psychological evaluation | Baseline, 3 month, 6 month and 12month follow-up assessments
  The Symptom Checklist - 90 (SCL-90) for evaluating general status, Self-Rating Depression Scale (SDS)for evaluating depression symptom,and Yale-Brown Obsessive Compulsive Scale (Y-BOCS) for evaluating obsessive compulsive symptom, will be utilized at each time point.
Personality evaluation | Baseline, 3 month, 6 month and 12month follow-up assessments
  The Eysenck Personality Questionnaire (EPQ)will be utilized at each time point.
Cognitive evaluation | Baseline, 3 month, 6 month and 12month follow-up assessments
  The Wechsler Memory Scale(WMS) for evaluating the memory will be utilized at each time point.
Evaluation of quality of life | Baseline, 3 month, 6 month and 12 month follow-up assessments
  The MOS item short from health survey(SF-36) be utilized at each time point.
Change in two static positron emission tomography(PET) images study | Baseline and 6month follow-up
  [18F]fluoro-D-glucose (FDG) for evaluating cerebral metabolism will be utilized at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Guo-dong Gao, M.D., Principal Investigator — Department of neurosurgery, Tangdu Hospital
Locations (1):
- Department of neurosurgery, Tangdu Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Chen L, Li N, Ge S, Lozano AM, Lee DJ, Yang C, Li L, Bai Q, Lu H, Wang J, Wang X, Li J, Jing J, Su M, Wei L, Wang X, Gao G. Long-term results after deep brain stimulation of nucleus accumbens and the anterior limb of the internal capsule for preventing heroin relapse: An open-label pilot study. Brain Stimul. 2019 Jan-Feb;12(1):175-183. doi: 10.1016/j.brs.2018.09.006. Epub 2018 Sep 14. PMID 30245163